CLINICAL TRIAL: NCT00818311
Title: Evaluation of the Effect of Photomodulation on Skin Safety Profile Following Different Schedules of Exposure to the Light Emitting Diode LED (Gentlewaves®) in Randomized Healthy Subjects
Brief Title: Skin Safety Profile of Different Exposure to the Light Emitting Diode (LED) in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Oreal (Industry)
Responsible Party: Dr Herndon / Dr Stephens, Thomas Stephens Associates 3310 Keller Springs Road Suite 130 Carrollton, TX 75006 USA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C08-D-121; 2008/US/LED/003
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Radiation Tolerance; Skin Aging; Rhytids
Keywords: Light emitting diode; tolerance; photomodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5 (Other)
  Interventions: Device: LED GentleWaves®

INTERVENTIONS:
Device: LED GentleWaves® — primary spectral radiance with a dominant 590 nm wavelength (yellow visible light), irradiance power level of 4mW/cm2, Light pulsed with sequential period on/off for a total duration of 35 seconds per cycle.
  Other Names: Gentle Waves professional base unit; The control unit consists of an LCD with the control electronics.; • primary spectral radiance with dominant 590 nm; • irradiance power level 4mW/cm2,; • Light pulsed with sequential period on/off for total duration of 35 seconds per cycle.

SUMMARY:
Photomodulation is a process which manipulates or regulates cell activity using light sources without thermal effect. Different studies have investigated the use of non-thermal low dose light emitting diode (LED) array for improving the appearance of photo aging damage. The photomodulation concept includes a low energy, narrow band or coherent light with specific pulse sequences and durations.

Preliminary investigations done by McDaniel et al. demonstrated that fibroblast activity could be regulated using pulsing light at specific wavelenghts. Using a variety of LED light sources, his group has demonstrated that by varying light pulses and other parameters, procollagen synthesis could be upregulated in human skin fibroblast culture [McDaniel DH, et al.Lasers Surg Med. 2002; 14-251]. A clinical correlation was also shown based on different clinical trials data on around 1000 subjects, LED has shown up to 90% improvement in wrinkles and an increase of collagen synthesis versus control with little or no side effects associated [Weiss, RA et al. Lasers Surg Med 2005; 36(2): 85-91- Weiss, RA et al.: J Drugs Dermatol 2004; 3(6): 605-610 - Weiss RA et al. Dermatol Surg 2005; 31(9):1999-1204 - Russel BA et al. J Cosmet Laser Ther 2005; 7 (3-4):196-200 - Bhat J et al. Laser Med Sci 2005; 20(1):6-10]. Based on these promising clinical data, Light BioScience submitted a dossier to the Food and Drug Administration (FDA) and obtained in January 2005 the FDA approval for its GentleWaves® Light Emitting Diode (LED) for the non-invasive treatment of periorbital (eye area) wrinkles and rhytids. The LED technology has been considered by FDA as non significant risk. In Europe, the GentleWaves® Light Emitting Diode has obtained the notified body certification for the same indication. This medical claim is associated with cosmetic improvement of aging and sun-damaged skin, further validation the science of LED photomodulation skin rejuvenation [Investigator's Brochure. Version 1].

This approval has been obtained with a professional LED GentleWaves® device used under a physician's responsibility. The initial regimen of 35 seconds twice per week with at least two days in between treatment for a total of 4 weeks duration of treatment has demonstrated efficacy for the treatment of typical signs of photo aging and no adverse effect.

A monocentre, randomized clinical study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate different treatment regimens in order to be able to develop new indications or to optimize the result already obtained in the treatment of wrinkles around the eyes. We therefore propose to perform a safety clinical trial with male and female volunteers with different schedules per day or per week.

A total of 100 subjects (male and female) will be randomized in the study according to the following schedule of exposure:

Group A: 20 subjects (8 males - 12 females) will be exposed to the LED twice a week for one cycle (35 seconds) with an interval between treatments of at least 2 days, during a treatment period of 4 weeks.

Group B: 20 subjects (8 males - 12 females) will be exposed to the LED twice a week for two consecutive cycles (35 seconds each) with an interval between treatments of at least 2 days, during a treatment period of 4 weeks.

Group C: 20 subjects (8 males - 12 females) will be exposed to the LED for one cycle (35 seconds) twice a day (morning and evening). This treatment will be repeated twice a week with an interval between treatments of at least 2 days, during a treatment period of 4 weeks.

Group D: 20 subjects (8 males - 12 females) will be exposed to the LED for one cycle (35 seconds) every day (from Monday to Friday) during a treatment of period of 4 weeks.

Group E: 20 subjects (8 males - 12 females) will be exposed to the LED for two consecutive cycles (35 seconds each) every day (from Monday to Friday) during a treatment of period of 4 weeks.

treatment period of 4 weeks.

Group D: 20 subjects (8 males - 12 females) will be exposed to the LED for one cycle (35 seconds) every day (from Monday to Friday) during a treatment of period of 4 weeks.

Group E: 20 subjects (8 males - 12 females) will be exposed to the LED for two consecutive cycles (35 seconds each) every day (from Monday to Friday) during a treatment of period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (male and female) at least 18 years old with skin types range from Fitzpatrick type I-VI (Appendix 1),
* Subjects must read, understand and sign the informed consent,
* Subjects must be willing and able to comply with follow up requirements,
* To be willing to report any medications taken during the study and refrain from taking any medication during the study that might produce photoreactions.

Exclusion Criteria:

* Subjects must not have active or localized or systemic infection,
* Subjects must not be immunocompromised,
* Subjects must be negative for HIV and hepatitis B and C serology,
* Subjects must not have history of light activated seizure or migraine headache disorder,
* Individuals taking medication who have been advised by a physician or pharmacist to avoid sunlight and subjects having vitiligo
* Subjects must not have mental illness such as schizophrenia or severe depression,
* Subjects must not have photosensitivity, photoallergy or photodermatitis,
* Subjects must not be pregnant or breast feeding. Subjects must discuss concerns about birth control with the study physician. Subjects who become pregnant during the study must inform the investigator immediately,
* Subject must not have a skin condition that the examining Investigator deems inappropriate for participation,
* Subject must not take part or intend to take part in another study liable to interfere with this study whatever the region of the body considered for 30 days prior to the study start and 30 days following completion of the study,
* Subjects must not have had GentleWaves treatment, other light treatments (including tanning beds), collagen or other facial tissue augmentation, Botox®, chemical peels, non-ablative (non invasive laser) therapies, dermabrasion, topical antioxidant or other resurfacing procedures at any time during the study,
* Subject must not refuse to sign the informed consent document and/or refuse to comply with all study requirements,
* Subjects must not have any previous history of keloïd scarring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assess the skin tolerance | 10

SECONDARY OUTCOMES:
Photography An overall global evaluation 2 biopsies | 10

CONTACTS AND LOCATIONS:
Overall Officials: James H Herndon, MD, Principal Investigator — Thomas Stephens and Associates, Inc
Locations (1):
- Thomas Stephens and Associates, Inc, Carrollton, Texas, United States